CLINICAL TRIAL: NCT04789876
Title: A Multicenter, Open-Label, Randomised Controlled Trial Investigating the Effectiveness Of The Phosphate Mobile App on Serum Phosphorus Outcomes In Adult Hemodialysis Patients With Hyperphosphatemia
Brief Title: Effectiveness of The Phosphate Mobile App on Serum Phosphorus in Adult Hemodialysis Patients With Hyperphosphatemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taylor's University (Other)
Responsible Party: Principal Investigator, Tilakavati Karupaiah, SRI Professor, Taylor's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEC 2019/011; NMRR-19-3825-45381 (Registry Identifier: National Medical Research Register)
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Hyperphosphatemia; End Stage Renal Disease on Dialysis
Keywords: Hemodialysis; Hyperphosphatemia; Mobile app; Dietary counseling; Serum phosphorus; Phosphate knowledge; Dietary intake; Phosphate binder adherence
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Intervention Model Description: Patients were allocated to the intervention and control group. The intervention group received a phosphate mobile app for 12 weeks and the control group received one-off dietary counselling delivered by a dietitian with a phosphate booklet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Intervention Group (AIG) (Experimental): Phosphate mobile app for 12 weeks.
  Interventions: Other: Phosphate mobile app
- Dietitian Intervention Group (DIG) (Active Comparator): One-off 45-minute dietary counselling delivered by a dietitian at the baseline of the study.
  Interventions: Behavioral: One-off dietary counselling with a phosphate booklet

INTERVENTIONS:
Other: Phosphate mobile app — The phosphate mobile app has the features of i) matching phosphate binder with dietary phosphate intake, ii) educational videos of phosphate management, iii) food database with local food items, iv) record-keeping and goal setting.
  Other Names: MyKidneyDiet - Phosphate Tracker
  Arms: App Intervention Group (AIG)
Behavioral: One-off dietary counselling with a phosphate booklet — One-off 45-minute dietary counselling delivered by a dietitian at the baseline of the study. Patients received a complimentary phosphate booklet after the counselling session. The phosphate booklet contains similar educational information as per the phosphate mobile app excluding the matching of phosphate binder with dietary phosphate information.
  Arms: Dietitian Intervention Group (DIG)

SUMMARY:
This multi-centred randomized, open label-controlled trial consists of hemodialysis (HD) patients identified with hyperphosphatemia (>1.78mmol/L). The intervention group received a phosphate mobile app and the control group received one-off dietary counselling for 12 weeks. Serum phosphate was measured pre-and post-intervention.

DETAILED DESCRIPTION:
This study is a multi-centred randomized, open label-controlled trial where a total of 66 HD patients (33 intervention vs 33 control) with hyperphosphatemia were recruited from government, private and non-governmental organization settings.

Patients who consented were subjected to screening for identification of hyperphosphatemia and other eligibility criteria. Patients who fulfilled the inclusion criteria were grouped according to shift and block randomized to either the intervention or control group using a web-based randomiser.

The intervention group received a phosphate mobile app for 12 weeks and the control group received one-off phosphate counselling delivered by a dietitian with a phosphate booklet. During the 12 weeks study period, patients in both control and intervention groups were assessed at baseline and 12 weeks for changes in serum phosphorus, serum corrected calcium, phosphate knowledge, dietary intake and phosphate binder adherence.

These parameters were compared at baseline and 12 weeks for within- and between-group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old and above.
* Patients were undergoing maintenance HD treatment for more than three months.
* Patients were on hemodialysis treatment for 4 hours per session, three times a week.
* Kt/V value (a numerical formula value to determine hemodialysis treatment adequacy. K is dialyser clearance of urea, t is dialysis time, and V is the volume of distribution of urea, approximately equal to the patient's total body water) is 1.2 and above each session.
* Patients were able to read English or Malay or Mandarin.
* Patients were on the single type of phosphate binder.
* Patients were having serum phosphorus above 1.78mmol/l and above for more than three months.
* Patients were not seen by a dietitian for the past one year for phosphate education.
* Patients did not have ward admission for the past three months.
* Patients did not have dementia or developmental delay.
* Patients owned and able to use a smartphone.
* Patients were able to use at least one comprehensive mobile application independently.
* Patients had access to the internet/data plan.
* Patients were willing to adhere to all study requirements and protocol.
* Patients were willing to accept the publication of data without exposing their name.

Exclusion Criteria:

* Patients were on incremental or acute hemodialysis.
* Patients had ward admission three months prior to the study and during the study period.
* Patients were terminally ill.
* Patients had cognitive impairment or physical disabilities (visual, hand dexterity, etc.) hindering interview and PMA utilisation.
* Patients had visual impairment or blind hindering the interview or the use of PMA.
* Patients were unable to self-care and dependent.
* Patients stayed in an institutionalised setting.
* Patients had undergone parathyroidectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Changes in serum phosphorus | Baseline, 12 weeks
  Effect of intervention on serum phosphorus

SECONDARY OUTCOMES:
Changes in phosphate knowledge | Baseline, 12 weeks
  A questionnaire used to assess phosphate knowledge and contained 18 questions related to phosphate treatment, disease pathophysiology, dialysis treatment, phosphate binder, dietary phosphate and responsibility. The questionnaire was an expert validated phosphate questionnaire with back-to-back-translation for English, Malay, and Chinese questionnaire. Each correct response was awarded 1 point, and all correct answers were summed to achieve a total score. The possible total score ranged from 0 to 18. All subjects completed this questionnaire at baseline and 12-week after the intervention.
Changes in dietary intake | Baseline, 12 weeks
  Dietary energy intake (kcal/day and kcal/kg body weight/day), dietary protein intake (g/day and g/kg body weight/day) and dietary phosphate (mg/day) assessed using a 3-day dietary record method at baseline and 12-week after the intervention.
Changes in phosphate binder adherence | Baseline, 12 weeks
  Phosphate binder adherence measured using the 4-item Morisky Medication Adherence Scale (MMAS) at baseline and 12-week after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tilakavati Karupaiah, PhD, Principal Investigator — Taylor's University; Teong Lee Fang, BSc, Study Chair — Taylor's University
Locations (3):
- Malaysia (3):
  - Pusat Rawatan Dialisis Islah, Batu Caves, Selangor
  - National Kidney Foundation Malaysia, Petaling Jaya, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ketteler M, Block GA, Evenepoel P, Fukagawa M, Herzog CA, McCann L, Moe SM, Shroff R, Tonelli MA, Toussaint ND, Vervloet MG, Leonard MB. Diagnosis, Evaluation, Prevention, and Treatment of Chronic Kidney Disease-Mineral and Bone Disorder: Synopsis of the Kidney Disease: Improving Global Outcomes 2017 Clinical Practice Guideline Update. Ann Intern Med. 2018 Mar 20;168(6):422-430. doi: 10.7326/M17-2640. Epub 2018 Feb 20. PMID 29459980
- [Background] Umeukeje EM, Mixon AS, Cavanaugh KL. Phosphate-control adherence in hemodialysis patients: current perspectives. Patient Prefer Adherence. 2018 Jul 4;12:1175-1191. doi: 10.2147/PPA.S145648. eCollection 2018. PMID 30013329
- [Result] Chan MW, Cheah HM, Mohd Padzil MB. Multidisciplinary education approach to optimize phosphate control among hemodialysis patients. Int J Clin Pharm. 2019 Oct;41(5):1282-1289. doi: 10.1007/s11096-019-00878-4. Epub 2019 Jul 13. PMID 31302884
- [Result] Milazi M, Bonner A, Douglas C. Effectiveness of educational or behavioral interventions on adherence to phosphate control in adults receiving hemodialysis: a systematic review. JBI Database System Rev Implement Rep. 2017 Apr;15(4):971-1010. doi: 10.11124/JBISRIR-2017-003360. PMID 28398983
- [Result] Fakih El Khoury C, Crutzen R, Schols JMGA, Halfens RJG, Karavetian M. A Dietary Mobile App for Patients Undergoing Hemodialysis: Prospective Pilot Study to Improve Dietary Intakes. J Med Internet Res. 2020 Jul 20;22(7):e17817. doi: 10.2196/17817. PMID 32706698
- [Result] Elder GJ, Malik A, Lambert K. Role of dietary phosphate restriction in chronic kidney disease. Nephrology (Carlton). 2018 Dec;23(12):1107-1115. doi: 10.1111/nep.13188. PMID 29064141
- [Result] Reddy V, Symes F, Sethi N, Scally AJ, Scott J, Mumtaz R, Stoves J. Dietitian-led education program to improve phosphate control in a single-center hemodialysis population. J Ren Nutr. 2009 Jul;19(4):314-20. doi: 10.1053/j.jrn.2008.11.001. PMID 19539185
- [Result] Vrdoljak I, Panjkota Krbavcic I, Bituh M, Leko N, Pavlovic D, Vrdoljak Margeta T. The impact of education and cooking methods on serum phosphate levels in patients on hemodialysis: 1-year study. Hemodial Int. 2017 Apr;21(2):256-264. doi: 10.1111/hdi.12468. Epub 2016 Aug 16. PMID 27528215